CLINICAL TRIAL: NCT00077935
Title: An Open-Label Multicenter Study Evaluating the Safety of Civamide Cream 0.075% as a Treatment in Subjects With Osteoarthritis of the Knee(s)
Brief Title: Civamide in OA of the Knee(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Study Director, Winston Laboratories, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WL-1001-05-04
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2004-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — zucapsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Civamide — Cream 0.075%, TID for 52 weeks

SUMMARY:
The purpose of this study is to evaluate the safety of Civamide Cream 0.075% as a Treatment in Subjects with Osteoarthritis (OA) of the Knee(s).

DETAILED DESCRIPTION:
This is a 52-week open label study wherein subjects are required to apply the study drug on the knee(s) three times a day. Subjects are required to return to the clinic every 13 weeks.

Enrollment Visit (Day 1) At the End-of-Study/Final Visit, Day 84 of Study No. WL-1001-05-01 (or preferably < 30 days following this visit) subjects will be invited to enroll in this long-term open label Study WL-1001-05-04. Subjects will sign a written informed consent prior to being enrolled into the long-term open label study. If enrolled at the final visit or < 30 days after the final visit of Study No. WL-1001-05-01, the final visit physical examination and laboratory examination will serve as baseline for this study. If enrolled > 30 days after the final visit, a new physical examination and laboratory examination will be completed upon enrollment into this study. The subjects will complete an OA Pain Score and Subject Global Evaluation (SGE) for their Target Knee, the same knee designated as the Target Knee in Study No. WL-1001-05-01. A 13-week supply of study drug and subject diaries for the next 13 weeks will be dispensed to each subject. Instructions on how to apply the study drug will be reviewed with the subjects. Subjects will also be instructed to complete their diaries daily (Adverse Events Log and Other Medications Log) and to return their completed diaries and study drug tubes at each clinic visit.

Treatment Period (Days 1- 365) Subjects will apply study drug to their Target Knee three times a day for 52 weeks. If the subject's other knee is affected by osteoarthritis pain, it may be treated with the study drug as well. The study drug tubes will be weighed prior to being dispensed to the subject. Each tube will also be weighed when the subject returns them.

At each clinic visit, the study staff will review the diaries with each subject for completeness and legibility.

Subjects will complete the OA Pain Score and Subject Global Evaluation at clinic visits on Day 1 and Weeks 13, 26, 39, and 52. Concurrent medications, adverse events, and study drug compliance will be reviewed and recorded by the study staff throughout the Treatment Period at clinic visits on Weeks 13, 26, 39, and 52 (End-of-Study/Final Visit). At the week 52 visit (End-of-Study/Final Visit), a physical examination and laboratory examination will be performed.

On Day 365 (End-of-Study/Final Visit) the subject will be discharged after all procedures have been completed.

ELIGIBILITY:
Inclusion Criteria

* Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent.
* Subject has participated (and not withdrawn secondary to any adverse event) in the Phase 3 Osteoarthritis Study WL-1001-05-01 and completed End-of-Study/Final Visit preferably < 30 days prior to Day 1 of this study (WL-1001-05-04).
* Subject is between 40 and 76 years of age.
* Subject is generally in good health.
* Subject is expected to be compliant with study procedures.
* Female subjects of child-bearing potential must have a negative urine pregnancy test at Day 1.
* Female subjects of child-bearing potential agree to use an approved form of contraception and must be on the same contraceptive method and dosage schedule during the entire study.

Exclusion Criteria

* Presence of tendonitis, bursitis, partial or complete joint replacement of knee(s).
* Presence of active skin disease, erythema, infection, wound, or irritation near the treatment area of the knee(s).
* Subject has an anticipated need for any surgical or other invasive procedure (e.g., synovial fluid aspiration, arthroscopy, tidal joint irrigation, injectable medications) that will be performed on the knees during the course of the study.
* Subject has a history and/or diagnosis of rheumatoid arthritis, fibromyalgia, connective tissue disease, psoriatic arthritis, erosive inflammatory OA, diffuse idiopathic skeletal hyperostosis, severe neurologic or vascular disease.
* Subject has active (redness, swelling, fever, etc.) gout or pseudo-gout within 6 months prior to screening.
* Subject has Type I or Type II diabetes with peripheral neuropathies.
* Subject has had trauma or surgery to the knee(s) within 1 year prior to the Enrollment Period.
* Subject has an underlying clinical condition, including previous malignancies that in the Investigator's judgment, is unstable.
* Subject has known allergy or hypersensitivity to capsicum, civamide, or capsaicin-containing products or any constituent of the cream formulation.
* Subject has a history of substance abuse within the past 12 months.
* Use of certain medications within the given restriction period prior to randomization and during the study.

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2003-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B. Phillips, M.D., Study Director — Winston Laboratories
Locations (34):
- United States (34):
  - Innovative Clinical Trials, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - OMC Clinical Research Center, Beverly Hills, California
  - Med. Investigations, Fair Oaks, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - Radiant Research, Daytona Beach, Florida
  - University Clinical Research, DeLand, Florida
  - Robert W. Levin, MD, Dunedin, Florida
  - University Clinical Research Inc., Pembroke Pines, Florida
  - Radiant Research, Atlanta, Georgia
  - Radiant Research, Boise, Idaho
  - Feinberg School of Medicine/Office of Clinical Rsrch and Trng, Chicago, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Chesapeake Medical Research, LLC, Baltimore, Maryland
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Medex Healthcare Research Inc., St Louis, Missouri
  - Arthritis Regional Research Center, Mercerville, New Jersey
  - New Mexico Research and Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Seligman Center for Advanced Therapeutics, New York, New York
  - NC Arthritis and Allergy Care Center, Raleigh, North Carolina
  - Raleigh Medical Group, PA, Raleigh, North Carolina
  - Piedmont Medical Group, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Beachwood, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Radiant Research, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Rheumatic Disease Associates, Ltd., Willow Grove, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Summit Research Solutions, Memphis, Tennessee
  - Radiant Research, Austin, Texas
  - Arthritis and Rheumatic Diseases, Portsmouth, Virginia
  - Physicians Pharmaceutical Study Services, Everett, Washington
  - Arthritis Clinic, Racine, Wisconsin